CLINICAL TRIAL: NCT04620070
Title: ON-SCENE Initiation of Extracorporeal CardioPulmonary Resuscitation (ECPR) During Refractory Out-of-Hospital Cardiac Arrest
Brief Title: ON-SCENE Initiation of Extracorporeal CardioPulmonary Resuscitation During Refractory Out-of-Hospital Cardiac Arrest
Acronym: ON-SCENE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Collaborators: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); Radboud University Medical Center (Other); University Medical Center Groningen (Other); Leiden University Medical Center (Other); Haga Hospital (Other); St. Antonius Hospital (Other); Isala (Other); Catharina Ziekenhuis Eindhoven (Other); Amphia ziekenhuis (Unknown)
Responsible Party: Principal Investigator, Dinis Reis Miranda, Principal Investigator, Erasmus Medical Center
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NL73073.078.20
Record Dates: First submitted 2020-10-26; First posted 2020-11-06 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Extracorporeal Membrane Oxygenation; Cardiac Arrest
Keywords: ECPR; prehospital ECPR; out of hospital cardiac arrest
MeSH Terms: conditions — Heart Arrest; Out-of-Hospital Cardiac Arrest

STUDY DESIGN:
Intervention Model Description: Stepped-wedge design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Conventional (No Intervention): In the Netherlands, out-of-hospital cardiac arrest (OHCA) is managed by paramedics. In this study, in the conventional arm, OHCA is managed by a physician of the Helicopter Emergency Medical Services (HEMS), but without the possibility of prehospital ECPR.
- Intervention group (Experimental): OHCA managed by the physician of the HEMS team, but with the possibility of prehospital ECPR.
  Interventions: Procedure: ECPR

INTERVENTIONS:
Procedure: ECPR — Application of prehospital ECPR
  Arms: Intervention group

SUMMARY:
Hypothesis: Implantation of on-scene ECPR by the HEMS teams in patients with sustained out-of-hospital cardiac arrest, results in the rapid return of circulation and, thus, improved survival and less neurological impairment, which is associated with lower health care costs.

DETAILED DESCRIPTION:
Rationale: Approximately half of all cardiac arrest patients achieve return of spontaneous circulation (ROSC) within 10 minutes. However, If ROSC is not achieved within 20 minutes, favourable neurological outcome is rare. Currently, patients without ROSC at scene die at scene, or are transported (while still in cardiac arrest) to the hospital. In the hospital, advanced life support is continued, or, when presented to selected hospitals capable for this strategy, patients receive Extracorporeal CardioPulmonary Resuscitation (ECPR). ECPR is a strategy in which a miniaturized heart-lung machine (similar to that used in open-heart surgery) is attached to the patient. Nowadays, the greatest drawback transporting OHCA patients with refractory arrest to the hospital are the low quality of thorax compression during transport and long time needed to arrive in the hospital, in part because not all hospitals are able to provide this treatment. In the Netherlands, Helicopter Emergency Medical Services (HEMS) deliver highly specialized medical care to trauma and non-trauma patients, covering the entire country.

Hypothesis: Implantation of on-scene ECPR by the HEMS teams in patients with sustained out-of-hospital cardiac arrest, results in the rapid return of circulation and, thus, improved survival and less neurological impairment, which is associated with lower health care costs.

Objective: To improve survival to hospital discharge and costs/QALY in young patients with OHCA by decreasing the time in cardiac arrest by initiating ECPR on scene.

ELIGIBILITY:
Inclusion Criteria:

* - Age between 18 and 50 years, known or as estimated at inclusion by the HEMS physician.
* Witnessed arrest (last seen well <5 min), OR signs of life (gasping, movement)
* Initial rhyme is VT/VF OR Suspected of having a pulmonary embolism
* Refractory cardiac arrest lasting longer than 20 minutes and shorter than 45 min

If age is not exactly known at inclusion and is estimated by the HEMS physician between 18 and 50 years but finally the patient appears to be younger or older, the patient will not be excluded.

Exclusion Criteria:

* - CO2 et<1.2 kPa (10 mmHg) during CPR
* No clear echographic visualisation of either the femoral artery or the femoral vein.
* Expected time from collapse to arrival at an ECPR center with a direct available ECPR team is less than 30 min.

The following patients will be withdrawn after initial inclusion as soon as the following information becomes available:

* Known malignancy
* Known intracranial haemorrhage/ischemia <6 weeks
* Care dependent for daily activities before arrest
* Patients with a "do not resuscitate" order, which was not known at time of the arrest.
* Refusal of deferred consent by the next of kin or by the patient himself to use the data. Deferred consent will not be asked to relatives of patients who die in scene, but are included in the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 221 (Actual)
Dates: Start 2021-10-15 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Hospital Survival | Hospital discharge (on average 6 weeks)
  (% patients surviving hospital discharge)

SECONDARY OUTCOMES:
Favourable neurological outcome (CPC 1-2) | 6 months after cardiac arrest
  (% of patients at least performing daily life activities independent)
Survival prehospital ECPR vs ECPR at the hospital vs no ECPR | Hospital discharge (on average 6 weeks after cardiac arrest)

CONTACTS AND LOCATIONS:
Overall Officials: Dinis Reis Miranda, Principal Investigator — Erasmus Medical Center
Locations (4):
- Netherlands (4):
  - Amsterdam UMC, Amsterdam
  - UMCG, Groningen
  - Radboud, Nijmegen
  - ErasmusMC, Rotterdam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ali S, Moors X, van Schuppen H, Mommers L, Weelink E, Meuwese CL, Kant M, van den Brule J, Kraemer CE, Vlaar APJ, Akin S, Lansink-Hartgring AO, Scholten E, Otterspoor L, de Metz J, Delnoij T, van Lieshout EMM, Houmes RJ, Hartog DD, Gommers D, Dos Reis Miranda D. A national multi centre pre-hospital ECPR stepped wedge study; design and rationale of the ON-SCENE study. Scand J Trauma Resusc Emerg Med. 2024 Apr 17;32(1):31. doi: 10.1186/s13049-024-01198-x. PMID 38632661